CLINICAL TRIAL: NCT07155252
Title: Home-based Oral Glucose Tolerance Test for Type 1 Diabetes Screening
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Breakthrough T1D (Other)
Responsible Party: Sponsor
Other Study IDs: 2000040441
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Single islet autoantibody: Participants with single islet autoantibody
  Interventions: Diagnostic Test: GTT@Home
- 2 or more positive islet antibodies: Participants with 2 or more positive islet antibodies who are in (Stage 1) or (Stage 2) without dysglycemia
  Interventions: Diagnostic Test: GTT@Home
- Recently diagnosed with diabetes: Participants meeting the diagnostic criteria for diabetes (stage 3 T1D) within 100 days from the diagnosis
  Interventions: Diagnostic Test: GTT@Home

INTERVENTIONS:
Diagnostic Test: GTT@Home — self-administered fingerstick based glucose tolerance test

SUMMARY:
This study aims at quantifying the accuracy of a self-administered fingerstick based glucose tolerance test (GTT@Home) respect to the gold-standard in-clinic venous plasma measures during the oral glucose tolerance test (OGTT) across a wide range of glycemic values in people at risk for clinical type 1 diabetes (T1D) (carriers of at least one islet autoantibody) or with new onset Stage 3 T1D within 100 days from the diagnosis.

DETAILED DESCRIPTION:
Investigators will conduct an observational longitudinal study that will include one home-based unsupervised GTT@Home test, a standard OGTT at a research facility and a supervised GTT@Home. Additionally, participants will have up to10-day blinded-CGM data collected.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥43 kg
* Presence of at least one islet autoantibody and/or≥ diagnosis of clinical T1D within 100 days.
* Documentation of the presence at least 1 islet autoantibody
* If participants meet ADA diagnostic criteria for Stage 3 type 1 diabetes, they will be eligible if the enrollment occurs within 100 days from the diagnosis and are at least 12 years old.
* Participants must be in good general health without other acute (e.g. infectious disease) febrile or chronic illnesses (e.g. uncontrolled asthma requiring high steroid doses, chronic arthritis) that in the judgment of the investigator could jeopardize participant safety or interfere with the study,
* Ability to give consent/assent
* Able to understand written and spoken English

Exclusion Criteria:

* Currently pregnant or becomes pregnant during the study
* Participants on sodium glucose cotransporter inhibitors (SGLTi).
* Donated blood in the past 8 weeks.

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 60 participants will be enrolled at the Yale University Pediatric and Adult Diabetes Clinic (New Haven, CT). To ensure there is wide variation in glucose ranges with glucose tolerance testing a total of 3 cohorts will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy of GTT@Home | up to 4 weeks from enrollment
  The accuracy will be quantified by correlation between GTT@Home and OGTT glucose measures as well as by the mean absolute relative difference between the two measures.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Galderisi, MD, Principal Investigator — Yale University
Locations (1):
- Yale University Pediatric and Adult Diabetes Clinic, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No